CLINICAL TRIAL: NCT02059317
Title: Evaluation of Dynamic Stability in the Low Back Pain Patient
Acronym: SDL
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2013/AD-02; 2013-A01379-36 (Other: ANSM)
Record Dates: First submitted 2014-02-06; First posted 2014-02-11 (Estimated); Last update posted 2025-11-19 (Actual); Status verified 2016-09

CONDITIONS: Low Back Pain; Chronic Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Rotation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Group 1: Six groups are created in order to randomized the order of interventions. In group 1, the order of interventions is as follows:
  1. Flexion-extension in the sagittal plane
  2. Rotation in a transverse plane
  3. Complex movement in three dimensions
  2 minutes of rest and walking occurs between interventions. The above-mentioned exercises (1, 2 & 3) are performed on day 0, day 7 and week 6 for patients, and only on day 0 for healthy volunteers.
  Interventions: Other: Flexion-extension in the sagittal plane; Other: Rotation in a transverse plane; Other: Complex movement in three dimensions
- Group 2: Six groups are created in order to randomized the order of interventions. In group 2, the order of interventions is as follows:
  1. Flexion-extension in the sagittal plane
  2. Complex movement in three dimensions
  3. Rotation in a transverse plane
  2 minutes of rest and walking occurs between interventions. The above-mentioned exercises (1, 2 & 3) are performed on day 0, day 7 and week 6 for patients, and only on day 0 for healthy volunteers.
  Interventions: Other: Flexion-extension in the sagittal plane; Other: Rotation in a transverse plane; Other: Complex movement in three dimensions
- Group 3: Six groups are created in order to randomized the order of interventions. In group 3, the order of interventions is as follows:
  1. Rotation in a transverse plane
  2. Flexion-extension in the sagittal plane
  3. Complex movement in three dimensions
  2 minutes of rest and walking occurs between interventions. The above-mentioned exercises (1, 2 & 3) are performed on day 0, day 7 and week 6 for patients, and only on day 0 for healthy volunteers.
  Interventions: Other: Flexion-extension in the sagittal plane; Other: Rotation in a transverse plane; Other: Complex movement in three dimensions
- Group 4: Six groups are created in order to randomized the order of interventions. In group 4, the order of interventions is as follows:
  1. Rotation in a transverse plane
  2. Complex movement in three dimensions
  3. Flexion-extension in the sagittal plane
  2 minutes of rest and walking occurs between interventions. The above-mentioned exercises (1, 2 & 3) are performed on day 0, day 7 and week 6 for patients, and only on day 0 for healthy volunteers.
  Interventions: Other: Flexion-extension in the sagittal plane; Other: Rotation in a transverse plane; Other: Complex movement in three dimensions
- Group 5: Six groups are created in order to randomized the order of interventions. In group 5, the order of interventions is as follows:
  1. Complex movement in three dimensions
  2. Flexion-extension in the sagittal plane
  3. Rotation in a transverse plane
  2 minutes of rest and walking occurs between interventions. The above-mentioned exercises (1, 2 & 3) are performed on day 0, day 7 and week 6 for patients, and only on day 0 for healthy volunteers.
  Interventions: Other: Flexion-extension in the sagittal plane; Other: Rotation in a transverse plane; Other: Complex movement in three dimensions
- Group 6: Six groups are created in order to randomized the order of interventions. In group 6, the order of interventions is as follows:
  1. Complex movement in three dimensions
  2. Rotation in a transverse plane
  3. Flexion-extension in the sagittal plane
  2 minutes of rest and walking occurs between interventions. The above-mentioned exercises (1, 2 & 3) are performed on day 0, day 7 and week 6 for patients, and only on day 0 for healthy volunteers.
  Interventions: Other: Flexion-extension in the sagittal plane; Other: Rotation in a transverse plane; Other: Complex movement in three dimensions

INTERVENTIONS:
Other: Flexion-extension in the sagittal plane — The movement required is a flexion - extension where the subject touches a target (adapted to his/her morphology) with both index fingers: the target is positioned in front of the subject, inline with his/her outstretched arms and at knee height. This movement simulates a lifting task without weight. The movement is repeated 30 times with a return to the initial position at a frequency of 0.32Hz.
Other: Rotation in a transverse plane — The movement required of the subject is a rotational movement where the subject alternately touches with his/her left and right hands two targets. The latter are positioned horizontally on either side of the subject at shoulder height and at arm's length. The movement is repeated 30 times at a frequency of 0.28 Hz.
Other: Complex movement in three dimensions — The subject is required to successively touch 4 targets situated (i) at knee height to the left of the subject, (ii) at shoulder height to the right of the subject, (iii) at shoulder height to the left of the patient, and (iv) at knee height to the right of the patient. The movement is repeated 30 times at a frequency of 0.16 Hz.

SUMMARY:
The main objective of this study is to compare on day 0 the maximum Lyapunov exponent (lmax, an indicator of local dynamic stability) of chronic low back pain patients versus that of healthy volunteers matched for age (± 5 years), sex and body mass index (BMI ± 15% of low back pain patients).

DETAILED DESCRIPTION:
The secondary objectives of this study are:

To compare lmax in the different experimental conditions within each group (chronic lower back pain patients, healthy volunteers).

To compare changes in lmax for low back pain patients at D7 and 6 weeks.

ELIGIBILITY:
General inclusion criteria:

* The patient/subject must have given his/her informed and signed consent
* The patient/subject must be insured or beneficiary of a health insurance plan

Inclusion criteria for low back pain patients:

* The patient has chronic low back pain lasting for more than 6 months and which is not postoperative in nature

General exclusion criteria:

* The patient/subject is participating in another study
* The patient/subject is in an exclusion period determined by a previous study
* The patient/subject is under judicial protection, under tutorship or curatorship
* The patient/subject refuses to sign the consent
* It is impossible to correctly inform the patient/subject
* The patient/subject is pregnant, parturient, or breastfeeding

Exclusion criteria for low back pain patients:

* The patient has a history of spinal surgery
* The patient has a history of preexisting postural disorder related to lumbalgia
* The patient has undergone a localized infiltration treatment (e.g. cortisone shots) in the last month
* The subject has a balance disorder, blindness, inability to carry out the experimental protocol

Exclusion criteria for healthy volunteers:

* The subject has a history of acute low back pain > 15 days or which has resulted in a work stoppage of more than 7 days in the 5 years preceding the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited during consultations in the department of Physical Medicine and Rehabilitation at the Nîmes University Hospital for lower back (lumbar) pain. The study population will include patients with chronic low back pain (lasting for more than 6 months and not postoperative).
  Healthy volunteers will be recruited at the Faculty of Medicine and the University Hospital of Nîmes.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2015-01; Primary Completion 2016-09-28 (Actual); Study Completion 2016-09-28 (Actual)

PRIMARY OUTCOMES:
the Lyapunov exponent (lmax, an indicator of local dynamic stability) | Day 0 (baseline)
  for flexion-extension movements
  The maximum Lyapunov exponent (lmax) is used to characterise local dynamic stability as in Rosenstein et al 1993 and Dingwell & Kang 2007.
the Lyapunov exponent (lmax, an indicator of local dynamic stability) | Day 0 (baseline)
  for rotational movements.
  The maximum Lyapunov exponent (lmax) is used to characterise local dynamic stability as in Rosenstein et al 1993 and Dingwell & Kang 2007.
the Lyapunov exponent (lmax, an indicator of local dynamic stability) | Day 0 (baseline)
  for complex movements.
  The maximum Lyapunov exponent (lmax) is used to characterise local dynamic stability as in Rosenstein et al 1993 and Dingwell & Kang 2007.

SECONDARY OUTCOMES:
the Lyapunov exponent (lmax, an indicator of local dynamic stability) | day 7
  for flexion-extension movements.
  The maximum Lyapunov exponent (lmax) is used to characterise local dynamic stability as in Rosenstein et al 1993 and Dingwell & Kang 2007.
the Lyapunov exponent (lmax, an indicator of local dynamic stability) | week 6
  for flexion-extension movements.
  The maximum Lyapunov exponent (lmax) is used to characterise local dynamic stability as in Rosenstein et al 1993 and Dingwell & Kang 2007.
the Lyapunov exponent (lmax, an indicator of local dynamic stability) | day 7
  for rotational movements.
  The maximum Lyapunov exponent (lmax) is used to characterise local dynamic stability as in Rosenstein et al 1993 and Dingwell & Kang 2007.
the Lyapunov exponent (lmax, an indicator of local dynamic stability) | week 6
  for rotational movements.
  The maximum Lyapunov exponent (lmax) is used to characterise local dynamic stability as in Rosenstein et al 1993 and Dingwell & Kang 2007.
the Lyapunov exponent (lmax, an indicator of local dynamic stability) | day 7
  for complex movements.
  The maximum Lyapunov exponent (lmax) is used to characterise local dynamic stability as in Rosenstein et al 1993 and Dingwell & Kang 2007.
the Lyapunov exponent (lmax, an indicator of local dynamic stability) | week 6
  for complex movements.
  The maximum Lyapunov exponent (lmax) is used to characterise local dynamic stability as in Rosenstein et al 1993 and Dingwell & Kang 2007.

OTHER OUTCOMES:
Sex | baseline (day 0)
  (male/female)
Age | baseline (day 0)
  (years)
weight (kg) | baseline (day 0)
Height (cm) | baseline (day 0)

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Dupeyron, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, France

REFERENCES:
- [Result] Graham RB, Dupeyron A, van Dieen JH. Between-day reliability of IMU-derived spine control metrics in patients with low back pain. J Biomech. 2020 Dec 2;113:110080. doi: 10.1016/j.jbiomech.2020.110080. Epub 2020 Oct 23. PMID 33157419